CLINICAL TRIAL: NCT06826508
Title: Modes of Delivery Impact Maternal Oxidative Stress Biomarkers and Dynamic Thiol Disulphide Homeostasis
Status: Completed | Type: Observational
Sponsor: Mardin Artuklu University (Other)
Collaborators: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Hasan Basri Savas, Associate Professor, Mardin Artuklu University
Other Study IDs: 18.09.2020 / 23-9
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Vaginal Delivery; Cesarian Section; Oxidative Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- vaginal delivery: 35 women who had spontaneous vaginal deliveries
- cesarean section: 23 women who had elective cesarean sections without labor

SUMMARY:
Modes of delivery impact maternal oxidative stress biomarkers and dynamic thiol disulphide homeostasis

ELIGIBILITY:
Inclusion Criteria:

For VD group:

* Women with spontaneous uncomplicated vaginal delivery
* Women who were in the 38th week and vertex presentation and whose contractions had started naturally.

For CS group:

• Women in their 38th week of pregnancy who delivered by elective CS without uterine contractions

Exclusion Criteria:

* Participants who were smokers
* Participants who had a non-optimal pre-pregnancy body mass index
* Systemic diseases such as diabetes mellitus and gestational hypertension.

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers | From January 2021 to August 2021
  Total antioxidation state (μmol Trolox equivalent/ L),
Oxidative stress markers | From January 2021 to August 2021
  Total oxidation status(μmol H2O2 equivalent/L)
Oxidative stress markers | From January 2021 to August 2021
  Oxidative stress index (arbitrary unit)
Oxidative stress markers | From January 2021 to August 2021
  Disulfide (-S-S-) (µmol / L) / alb (g / l)
Oxidative stress markers | From January 2021 to August 2021
  Total thiol (µmol / L)
Oxidative stress markers | From January 2021 to August 2021
  Native thiol (µmol / L) / alb (g / l)
Oxidative stress markers | From January 2021 to August 2021
  Ischemia modified albumin (U/L)
Oxidative stress markers | From January 2021 to August 2021
  Paroxanase (U/L)
Oxidative stress markers | From January 2021 to August 2021
  Arylesterase (Ku/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Training and Research Hospital Gynecology and Obstetrics Department, Antalya, Turkey (Türkiye)